CLINICAL TRIAL: NCT04824079
Title: Study of Keynatinib in Patients With Advanced Non-small Cell Lung Cancer With Brain Metastasis or Progression of Brain Metastasis After Treatment With EGFR Inhibitor(s)
Brief Title: Keynatinib in Treated Patients With NSCLC and Brain Metastases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medolution Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEDO-007-20002
Record Dates: First submitted 2021-03-23; First posted 2021-04-01 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Non-Small Cell Lung Cancer With EGFR Mutation; Brain Metastases
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Keynatinib treatment group (Experimental): All subjects shall be treated with Keynatinib twice a day (once every 12±3 hours), 20 mg each time, fasting within 2 hours before and 1 hour after taking the drug, and taking warm water when taking the drug. Every 21 days is a treatment cycle .
  Interventions: Drug: Keynatinib

INTERVENTIONS:
Drug: Keynatinib — The recommended dose is 20 mg Keynatinib twice a day until disease progression， unacceptable toxicity death occurs or withdraw from the study, whichever occurs first.
  Other Names: TL007

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Keynatinib capsules in patients with advanced non-small cell lung cancer (NSCLC) with brain metastasis or progression of brain metastasis after treatment with EGFR inhibitors. As well as, to evaluate the penetration rate of Keynatinib in the Blood-Brain Barrier (BBB) and its PK characteristics, and the relationship between exposure levels with efficacy and safety.

DETAILED DESCRIPTION:
This is a multicenter, non-randomized, open, single-arm, phase IIa trial investigating the security and effectiveness of Keynatinib in patients with advanced non-small cell lung cancer (NSCLC) with brain metastasis or progression of brain metastasis after treatment with EGFR inhibitors.

ELIGIBILITY:
Inclusion Criteria:

1. Unlimited gender, age ≥ 18 years；
2. Histologically or cytologically documented locally advanced, metastatic NSCLC (including L858R and/or Exon19 del mutation positive). The EGFR mutation assessed by local laboratory/or central laboratory via tissue/cytology or in plasma;
3. Subjects should have the following conditions: a. (Cohort 1) Progression on any of the first or second generation EGFR inhibitors (gefitinib, erlotinib, afatinib, etc.).B. (Cohort 2) Progression on any third generation EGFR inhibitor (oxitinib, etc.), prior or non-prior treatment with any first or second generation EGFR inhibitor;
4. The peripheral lesions did not progress after EGFR inhibitor treatment, but the occurrence of brain metastasis or progression of brain metastasis was confirmed by magnetic resonance imaging (MRI);
5. As determined by the investigator, no final surgical resection or radiotherapy is expected for all lesions;
6. Stable condition for at least 2 weeks prior to study medication without any corticosteroid or anticonvulsant therapy;
7. The status score of Eastern Cooperative Oncology Group (ECOG) is 0 to 1 points, and there was no deterioration during the first 2 weeks of enrollment;
8. Estimated survival time > 3 months；
9. Sufficient bone marrow, liver, kidney and blood coagulation function；
10. Subjects must be willing to use barrier contraception；
11. Ability to provide informed consent, complete all study assessments and have complete medical record.

Exclusion Criteria:

1. Have previously received chemotherapy, immunotherapy or any other systemic antitumor therapies within 4 weeks before the first administration; Have previously received EGFR-TKI within 5× half-life before the first administration; Have received oral fluorouracil and other small-molecule targeted drugs (whichever is longer) within 2 weeks or 5× half-life before enrollment; Within 2 weeks before enrollment, subjects had received palliative radiotherapy for non-target lesions for symptom relief, and traditional Chinese medicine (including Chinese patent medicine) for tumor indication;
2. Have received whole brain radiation therapy;
3. Only leptomeningeal metastasis are present;
4. Historical intracranial hemorrhage not related to the tumor;
5. Major organ surgery (excluding needle biopsy) or significant trauma have been performed within 4 weeks prior to enrollment;
6. The drug or food with strong inhibition or induction of cytochrome P450 (CYP) isoenzyme CYP3A4 could not be stopped. The drug or food with strong inhibition or induction of cytochrome P450 (CYP) isoenzyme CYP3A4 had been used within 7 days before enrollment;
7. Any unresolved toxicities from prior therapy greater than CTCAE 5.0 grade 1 at the time of enrollment with the exception of alopecia;
8. Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the tablet or previous significant bowel resection that would preclude adequate absorption of Keynatinib;
9. Past medical history of ILD, drug-induced ILD, radiation pneumonitis which required steroid treatment, or CT scan at baseline revealed the presence of idiopathic pulmonary fibrosis; Uncontrolled large pleural effusion or pericardial effusion; Active tuberculosis;
10. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses or active infection including hepatitis B, hepatitis C and HIV;
11. Have a history of severe cardiovascular disease (NYHA cardiac function grade III or IV);
12. Other primary malignancies (except cured basal cell carcinoma of the skin and carcinoma in situ of the cervix) within 5 years;
13. Allergic to the active ingredient or excipient of Keynatinib;
14. Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-10-21 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate | From start of treatment to time of progression (in CNS or non-CNS disease) , intolerable toxicity, withdrawal of informed consent or death, whichever occurs first，assessed up to 2 years.
  The proportion of subjects whose optimal efficacy observed from the beginning of administration is CR or PR.

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Shandong Cancer Hospital, Jinan, Shandong

IPD SHARING:
Plan to Share IPD: No